CLINICAL TRIAL: NCT05167084
Title: Acute Consequences Of Food-induced Glucocorticoid Secretion In Healthy Individuals - A Double-blind, Randomized, Placebo-controlled Cross-over Study
Brief Title: Acute Consequences Of Food-induced Glucocorticoid Secretion In Healthy Individuals
Acronym: Gluco-Feed
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eleonora Seelig (Other)
Responsible Party: Sponsor-Investigator, Eleonora Seelig, Principal Investigator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EKNZ 2021-01507
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Glucocorticoid Effect
Keywords: cortisol; overfeeding; glucocorticoids; insulin sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Metyrapone

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled cross-over study
Who Masked: Participant, Investigator
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metyrapone And Hydrocortisone (Experimental): During one of the study periods, subjects receive hydrocortisone 19.9 mg/d subcutaneously via a pump in a pulsed fashion (eight times/day) and metyrapone per os (starting with a dose of 500 mg/d, then the dose will be increased the next days until 2500mg/d is achieved).
  Interventions: Drug: Metyrapone 250 mg Oral Tablets; Drug: Hydrocortisone 19,9mg s.c., pulsatile with a flow rate of 10μl/s
- Placebo (Placebo Comparator): During the other study period, subjects receive placebo (0,9% NaCl solution) 19.9 mg/d subcutaneously via a pump in a pulsed fashion and the same dose of placebo tablets p.o instead of metyrapone.
  Interventions: Drug: Placebo 250 mg Tablets; Drug: Placebo (0,9% NaCl solution)

INTERVENTIONS:
Drug: Metyrapone 250 mg Oral Tablets — During one phase of the study: Metyrapone (pills of 250mg) on full stomach: Day 1 0-1-1, day 2 1-2-2, day 3 2-2-3 day 4 3-3-4 day 5 3-3-4 day 6 3-3-4 day 7 3-3-4 day 8 3-0-0
  Arms: Metyrapone And Hydrocortisone
Drug: Placebo 250 mg Tablets — During another phase of the study: identical looking placebo pills starting Day 1 0-1-1, day 2 1-2-2, day 3 2-2-3 day 4 3-3-4 day 5 3-3-4 day 6 3-3-4 day 7 3-3-4 day 8 3-0-0
  Arms: Placebo
Drug: Hydrocortisone 19,9mg s.c., pulsatile with a flow rate of 10μl/s — Hydrocortisone will be delivered subcutaneously via a pump in a pulsed fashion with a flow rate of 10μl/s from day 1 to day 8 in a total daily dose of 19.9mg
  Arms: Metyrapone And Hydrocortisone
Drug: Placebo (0,9% NaCl solution) — Placebo (0,9% NaCl solution) 19.9 mg/d subcutaneously via a pump in a pulsed fashion with a flow rate of 10μl/s from day 1 to day 8
  Arms: Placebo

SUMMARY:
In a randomized, cross-over study, 20 healthy volunteers will receive a block and replace therapy that mimics physiological GC rhythm (metyrapone plus hydrocortisone) or placebo. Participants will undergo two identical overfeeding periods with each treatment. With the block and replace therapy, food-induced GC peak will be suppressed. Metabolic and autonomic parameters will be compared to reveal, whether GCs mediate the physiological adaptions to excessive food intake.

Understanding acute effects of GCs upon food intake is critical, since repetitive disruptions of GC secretion may become harmful in chronic conditions.

DETAILED DESCRIPTION:
Obesity is one of the most serious health problems of the 21st century. To understand how we regulate our body weight is crucial for developing new treatment targets. Even though body mass index of populations is increasing, the body weight of adults is usually kept stable over time. Indeed, acute excessive food intake triggers a set of adaptions in order to prevent weight gain. The signal that triggers these beneficial adaptions is still unknown. Glucocorticoid (GC) secretion increases with acute food intake and many physiological adaptions to overfeeding coincide with classical glucocorticoid actions. The investigators therefore hypothesize that GCs are the signal that prevents weight gain during acute overfeeding.

The objective of this project is to test whether food-induced GCs represent the physiological signal that defends against weight gain.

The primary objective is to investigate whether reduction in insulin sensitivity is abolished with the block and replace therapy.

Secondary objectives are to investigate whether suppression of GC secretion during excessive food intake impairs the activation of sympathetic nervous system, satiety, satiation, energy expenditure, substrate utilization, blood pressure, secretion of neuroendocrine hormones, lipids and immune cells.

This is a double-blind, randomized, placebo-controlled cross-over study. After screening, subjects will be randomized to two crossover 8-day study periods with a washout period of 28 days:

A) Participants will receive hydrocortisone 19.9 mg/d subcutaneously via a pump in a pulsed fashion (eight times/day) and metyrapone per os (starting with a dose of 500 mg/d on day 1 to 2500mg/d on day 4, and then will be kept constant until day 8)

B) Participants will receive placebo (0,9% NaCl solution) 19.9 mg/d subcutaneously via a pump in a pulsed fashion and placebo pills per os (starting with a dose of 500 mg/d on day 1 to 2500mg/d on day 4, and then will be kept constant until day 8)

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 25 kg/m2

Exclusion Criteria:

* Previous medical history for any chronic condition in the last three months, active disease or abnormal physical examination as verified by a qualified physician.
* Casual smoking (>6 cigarettes per day)
* Frequent, heavy alcohol consumption (>30g/day)
* Frequent, heavy caffeine consumption (>4 caffeinated drinks/day)
* Regular physical exercise (>4hrs per week)
* Shift workers
* Participation in an investigational drug trail within the past two months
* Intake of any drugs (prescribed, over the counter or recreational) including topical steroids and inhalers, within 48 hours of the study initiation
* Known allergy to metyrapone
* Inability or unwillingness to provide informed consent

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since hormone fluctuations associated with the menstrual cycle may alter cortisol levels, women will not be included in the study. Although diversity will be reduced and the statements of the study cannot be applied to the female sex, these strict inclusion criteria allow an optimal homogeneity and increase statistical power.
Enrollment: 20 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Two 8-day intervention periods
  Change in insulin sensitivity assessed with a mixed meal tolerance test

SECONDARY OUTCOMES:
Cortisol (nmol/l) total and free | Two 8-day intervention periods
  Blood sample
Renin | Two 8-day intervention periods
  Blood Sample
Aldosterone (Adrenal Steroid Hormones) | Two 8-day intervention periods
  Blood Sample
Pregnenolon (Adrenal Steroid Hormones) | Two 8-day intervention periods
  Blood Sample
Progesteron (Adrenal Steroid Hormones) | Two 8-day intervention periods
  Blood Sample
11-Deoxycorticosteron (Adrenal Steroid Hormones) | Two 8-day intervention periods
  Blood Sample
Corticosteron (Adrenal Steroid Hormones) | Two 8-day intervention periods
  Blood Sample
18-Hydroxycorticosteron (Adrenal Steroid Hormones) | Two 8-day intervention periods
  Blood Sample
17-Hydroxypregnenolon (Adrenal Steroid Hormones) | Two 8-day intervention periods
  Blood Sample
17-Hydroxyprogesteron (Adrenal Steroid Hormones) | Two 8-day intervention periods
  Blood Sample
11-Deoxycortisol (Adrenal Steroid Hormones) | Two 8-day intervention periods
  Blood Sample
GLP-1 (nmol/l) | Two 8-day intervention periods
  Blood sample
GIP (nmol/l) | Two 8-day intervention periods
  Blood Sample
PYY (pg/ml) | Two 8-day intervention periods
  Blood Sample
T3 (nmol/l) | Two 8-day intervention periods
  Blood Sample
T4 (nmol/l) | Two 8-day intervention periods
  Blood Sample
TSH (mIU/l) | Two 8-day intervention periods
  Blood Sample
HGH (mIU/l) | Two 8-day intervention periods
  Blood Sample
Lipids (mmol/l) ((total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides) | Two 8-day intervention periods
  Blood Sample
GDF-15 (pg/mL) | Two 8-day intervention periods
  Blood Sample
Sympathetic nervous system activity | Two 8-day intervention periods
  Heart rate variability analysis
Systolic and diastolic blood pressure | Two 8-day intervention periods
  Assessment of blood pressure with a standard blood pressure monitor.
Weight | Two 8-day intervention periods
  Measurement of weight with a standard scale
Energy expenditure | Two 8-day intervention periods
  Basal metabolic rate measured with indirect calorimetry
Substrate utilisation | Two 8-day intervention periods
  Respiratory quotient assessed with indirect calorimetry
Satiety | Two 8-day intervention periods
  Appetite rating with visual analogue scale (VAS) from 0mm-100mm (0mm=not at all and 100mm=extreme)
Satiation | Two 8-day intervention periods
  Amount of food intake with ad libitum buffet

OTHER OUTCOMES:
IL-6 (Inflammatory markers) | Two 8-day intervention periods
  Blood Sample
IL-1RA (Inflammatory markers) | Two 8-day intervention periods
  Blood Sample
IL-8 (Inflammatory markers) | Two 8-day intervention periods
  Blood Sample
CRP (Inflammatory markers) | Two 8-day intervention periods
  Blood Sample
Metabolomics | Two 8-day intervention periods
  Metabolomics will be performed in blood plasma

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No